CLINICAL TRIAL: NCT05477810
Title: Single-center, Open-label, Randomized, Two-period, Two-way Crossover Study to Investigate the Bioequivalence of a Single-dose of 12 mg IVERMECTIN Administered as Orally Disintegrating Mini Tablets (CHILD-IVITAB) Versus a Single-dose of 12 mg Regular IVERMECTIN Tablets (STROMECTOL) in Healthy Adults Under Fasting Conditions
Brief Title: Bioequivalence of a Single-dose of 12 mg IVERMECTIN as Orally Disintegrating Mini Tablets Versus a Single-dose of 12 mg Regular IVERMECTIN Tablets in Healthy Adults Under Fasting Conditions
Acronym: CHILD-IVITAB
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Permamed AG, Switzerland (Unknown); Galvita AG, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2022-01276; ks21Pfister2
Record Dates: First submitted 2022-07-20; First posted 2022-07-28 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Bioequivalence
Keywords: CHILD-IVITAB; STROMECTOL; Ivermectin; Palatability
MeSH Terms: interventions — Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: open-label, randomized, two-period, two-way crossover, single-dose bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (CHILD-IVITAB) before Treatment B (STROMECTOL) (Experimental): A single oral dose of 12 mg CHILD-IVITAB administered as four ODTs of 3 mg (given in the fasted state in the morning).
  A single oral dose of 12 mg STROMECTOL administered as four tablets of 3 mg (given in the fasted state in the morning).
  The wash-out period between doses will be at least 7 days.
  Interventions: Drug: Treatment A (investigational drug) followed by Treatment B (reference drug); Drug: Treatment B (reference drug) followed by Treatment A (investigational drug)
- Treatment B (STROMECTOL) before Treatment A (CHILD-IVITAB) (Active Comparator): A single oral dose of 12 mg STROMECTOL administered as four tablets of 3 mg (given in the fasted state in the morning).
  A single oral dose of 12 mg CHILD-IVITAB administered as four ODTs of 3 mg (given in the fasted state in the morning).
  The wash-out period between doses will be at least 7 days.
  Interventions: Drug: Treatment A (investigational drug) followed by Treatment B (reference drug); Drug: Treatment B (reference drug) followed by Treatment A (investigational drug)

INTERVENTIONS:
Drug: Treatment A (investigational drug) followed by Treatment B (reference drug) — Two drug administration periods (1 and 2), each consisting of administration of Treatment A (investigational drug) followed by Treatment B (reference drug) on Day 1 will be performed. Post administration of the study drug standard PK sampling, measurement of vital signs, adverse events, ECG and VAS as per schedule will be done over a time period of 11 hours. The study participants will thereafter be discharged. The participants will return to the study center at 24, 48, 72 and 96 hours after study drug administration in each treatment period for blood sampling, vital signs and safety assessments as per schedule. The wash-out period between doses will be at least 7 days.
Drug: Treatment B (reference drug) followed by Treatment A (investigational drug) — Two drug administration periods (1 and 2), each consisting of administration of Treatment B (reference drug) followed by Treatment A (investigational drug) or on Day 1 will be performed. Post administration of the study drug standard PK sampling, measurement of vital signs, adverse events, ECG and VAS as per schedule will be done over a time period of 11 hours. The study participants will thereafter be discharged. The participants will return to the study center at 24, 48, 72 and 96 hours after study drug administration in each treatment period for blood sampling, vital signs and safety assessments as per schedule. The wash-out period between doses will be at least 7 days.

SUMMARY:
This is a phase I, single-center, open-label, randomized, two-period, two-way crossover, single-dose bioequivalence study in which the active substance ivermectin is administered as a single dose of 12 mg as either CHILD-IVITAB or STROMECTOL during two study drug administration periods. Each treatment will be investigated in the same subgroup of 16 healthy male or female study participants under fasted conditions.

DETAILED DESCRIPTION:
Ivermectin is used in humans as an oral antiparasitic agent. Currently approved ivermectin tablets are designed for adult patients. A child-appropriate formulation is not yet available. Ivermectin in suspension is not practicable as the stability is fragile, the shelf-life is very short, and the suspension is affected by UV light exposure. If tablets are offered to infants and young children as crushed or in a suspended form they are prone to imprecise dosing (loss of product after crushing or sedimentation of product after suspension). They are not palatable, and thereby frequently expelled out of the mouth by the child. All above compromise drug-adherence and effectiveness of treatment. In this bioequivalence study in healthy adults, CHILD-IVITAB, a novel orally disintegrating tablet (ODT) formulation containing the active ingredient ivermectin, will be evaluated. CHILD-IVITABs are stable in hot and humid atmosphere and no external agent is required for taste masking or swallowing. This study aims to determine if 12 mg of CHILD-IVITAB administered in a single dose is bioequivalent (with 0.80, 1.25 as the bioequivalence boundaries for AUC0-∞) to 12 mg administered as a single dose of the reference formulation STROMECTOL under fasting conditions. Further this study aims to characterize tolerability of CHILD-IVITAB in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 45 years (inclusive) at screening.
* Healthy adult females on contraceptives at least 1 month prior to the start of the study until 1 month after the completion of the study and urine pregnancy test at screening and pre-study drug administration negative.
* No history of alcohol or drug abuse.
* No history of chronic liver or kidney disease.
* No clinically significant findings on the physical examination at screening.
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive) at screening.
* Normal blood pressure and heart rate (Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and heart rate (HR) 45-90 bpm (inclusive), measured after 5 minutes in the supine position at screening).
* Hematology and blood chemistry results not deviating from the normal range to a clinically relevant extent at screening. Gilbert's syndrome (increased total and unconjugated bilirubin when fasting) will be accepted if mild.
* A 12-lead ECG without significant abnormalities (QTc ³450 msec at screening or pronounced sinus bradycardia (<40 bpm/min), even if elicited by sport)
* Negative urine drug screen (amphetamines, benzodiazepines, cannabis, cocaine, and opiates).
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.
* The participant agrees to be available for scheduled visits.
* Informed and signed consent obtained prior to any study-mandated procedure (including specific request for HIV serology and hepatitis as well as for urinary screen for drugs).

Exclusion Criteria:

* Eligible participants must meet none of the following exclusion criteria:
* Known hypersensitivity to any excipients of the drug formulations.
* Treatment with another investigational drug within 3 months prior to screening.
* Participation in a clinical study/trial in the previous 3 months unless no treatment taken or large amounts of blood collected
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Significant caffeine consumption defined as > 400 mg per day at screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* History of moderate or severe allergy or asthma at any time. Allergic rhinitis is acceptable if non symptomatic when starting the study and if symptoms are not anticipated to occur during the first 4 weeks of each period and are not expected to require a corticosteroid treatment.
* History of cardiovascular dysfunction if considered as clinically relevant (conduction abnormality, arrhythmia, bradycardia, angina pectoris, cardiac hypertrophy unless elicited by training, embolism).
* Recurrent hypotensive events considered as clinically relevant.
* Intense sport activities up to 4 days before inclusion
* Use of any medication the week prior to study or as based on 5 plasma half-life rule (before screening, after screening) and throughout study. Paracetamol is permissible before the study as a rescue medication but only with investigator's permission.
* Smoking (consumption of ≤5 cigarettes/day or equivalent is acceptable, provided the subject commits to quit entirely during the study)
* Loss of 350 ml or more of blood or blood donation within 3 months prior to screening.
* Positive results from the hepatitis serology, except for vaccinated (hepatitis B virus) participants, at screening.
* Positive results from the HIV serology at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening. l

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics (PK) primary endpoint | At Baseline, at 30 and 60 minutes, at 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours after study drug administration in each treatment period
  Change in the area under the plasma concentration-time curve from zero to infinity (AUC0-∞) of ivermectin in each treatment period

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) of ivermectin in each treatment period | Over a time period of 11 hours after study drug administration in each treatment period
  The maximum plasma concentration (Cmax) of ivermectin in each treatment period
The area under the plasma concentration-time curve from time zero to time t of the last measured concentration above the limit of quantification (AUC0-tlast) of ivermectin in each treatment period | Over a time period of 11 hours after study drug administration in each treatment period
  The area under the plasma concentration-time curve from time zero to time t of the last measured concentration above the limit of quantification (AUC0-tlast) of ivermectin in each treatment period
The time to reach maximum plasma concentration (tmax) of ivermectin in each treatment period | Over a time period of 11 hours after study drug administration in each treatment period
  The time to reach maximum plasma concentration (tmax) of ivermectin in each treatment period
Supine blood pressure (systolic and diastolic) | At Baseline, at 2, 4, 24, 48, 72 and 96 hours after study drug administration in each treatment period and at Day 7-10 of period 2
  Change from baseline to each time point of measurement during each treatment period as per study schedule for supine blood pressure
ECG (conduction changes) | At Baseline, at 2, 4 hours after study drug administration in each treatment period and at Day 7-10 of period 2
  Change from baseline to each time point of measurement during each treatment period as per study schedule for ECG variables (conduction system)
Adverse events (AEs) reporting from first drug administration up to end of study (EOS) (number of AEs) | From Baseline until Day 7-10 of period 2 (between 4 to a maximum of 7 weeks)
  Adverse events (AEs) reporting from first drug administration up to EOS
Tolerability of Treatments A and B utilizing a visual analogue scale (VAS) for gastrointestinal tract (GIT) (2 items) | At Baseline, at 30 and 60 minutes, at 2, 3, 4, 6, 10 hours after study drug administration in each treatment period
  Tolerability of Treatments A and B utilizing a VAS for GIT (2 items) ; (0 = tolerable; 10 = very untolerable)
Tolerability of Treatments A and B utilizing a VAS for central nervous system (CNS) (6 items) | At Baseline, at 30 and 60 minutes, at 2, 3, 4, 6, 10 hours after study drug administration in each treatment period
  Tolerability of Treatments A and B utilizing a VAS for CNS (6 items); (0 = tolerable; 10 = very untolerable)
Palatability of Treatments A and B utilizing a VAS (bitterness, sweetness, intensity, and palatability/acceptability) | At 0 and at 30 minutes after study drug administration in each treatment period
  Palatability of Treatments A and B utilizing a VAS (bitterness, sweetness, intensity, and palatability/acceptability); (0 = pleasant; 10 = very unpleasant)
Heart rate | At Baseline, at 2, 4, 24, 48, 72 and 96 hours after study drug administration in each treatment period and at Day 7-10 of period 2
  Change from baseline to each time point of measurement during each treatment period as per study schedule for Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pfister, Prof. Dr. med., Study Director — Universitäts-Kinderspital beider Basel (UKBB); Laura Rothuizen, Dr. med., Principal Investigator — University Hospital CHUV, Service of Clinical Pharmacology
Locations (1):
- University Hospital CHUV, Service of Clinical Pharmacology, Lausanne, Switzerland